CLINICAL TRIAL: NCT05488418
Title: Étude Clinique Des Biomarqueurs de la résilience au Stress: rôle d'ELK1 et GPR56
Brief Title: Clinical Study of Biomarkers of Stress Resilience: Role of ELK1 and GPR56
Acronym: GeBra-clin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM21_0492; ID-RCB (Other: 2022-A00070-43)
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Anxiety Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients exposed to a potentially traumatic event (Experimental)
  Interventions: Other: Clinical, cognitive and biological tests

INTERVENTIONS:
Other: Clinical, cognitive and biological tests — Evaluations at 1, 3, 6 and 12 months post-inclusion will be performed, during which the subject will complete various clinical and cognitive tests.
  A blood sample will be collected at each visit to study biological processes including the regulation of genetic and epigenetic expression, in particular the expression of the GPR56 and ELK1 genes in the blood.
  For eligible subjects a brain MRI will be proposed at the first visit.
  Other Names: Blood sample collection; Cerebral MRI exam

SUMMARY:
70% of Europeans will be exposed to a potentially traumatic event (PTE). Following this experience, people are likely to develop various psychiatric disorders such as post-traumatic stress disorder (PTSD) or a major depressive episode (MDE). However, not all subjects have the same risk to develop a pathology, and resilience capacities, which depend on multiple factors are difficult to predict. Currently, there are no objective tools to stratify exposed subjects according to their risk of developing pathological responses to stress, which leads to difficulties in allocating means of prevention and treatment.

Recently, new biological hypotheses explaining vulnerability/resilience to stress and depression, implicating the GPR56 and ELK1 genes, have been described. Previous studies have shown that evaluation of the vulnerability risk can be obtained from clinical, cognitive, biological or brain imaging variables, but no study has integrated these different approaches. Therefore, the project presented here aims at integrating behavioral, biological and neuroimaging data to predict the development of psychiatric disease. In this study, a prospective cohort of 255 violent trauma victims will be set up in 3 French cities for a period of 2 years. Eligible subjects will be included in the month following PTE and will be followed longitudinally for 12 months. Evaluations at 1, 3, 6 and 12 months will be performed, during which the subject will complete various clinical and cognitive tests. A blood sample will be collected at each visit to study biological processes including the regulation of genetic and epigenetic expression, in particular the expression of the GPR56 and ELK1 genes in the blood. For eligible subjects a brain MRI will be proposed at the first visit.

We hypothesize that the genetic expression of ELK1 and GPR56 is predictive of the development of psychiatric pathologies at 6 and 12 months post-PTE. The ambition of this project is also to highlight the importance of a multimodal approach integrating a triad of markers (behavioral, biological and neuroimaging) to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to a traumatic event within 30 days, as defined by ESA criteria A of the DSM-5
* Signed free and informed consent
* Covered by a health insurance company
* 18 to 65 years at inclusion
* Available for a 12-month period follow-up
* Have the ability to speak, read, and understand French
* Have the ability to complete clinical evaluations and self-report measures at baseline and throughout the study

Exclusion Criteria:

* Have any condition for which, in the opinion of the investigator or designee, study participation would not be in their best interest (including but not limited to unstable general medical condition, pregnancy) or that could prevent, limit, or confound the protocol-specified assessments
* One or more criteria for ineligibility for registration on the National Registry of Volunteers for Research Involving Humans (VRB)
* History of stable or non-stable psychiatric illness such as bipolar disorder or schizophrenia or any other pathology that may interfere with the evaluations
* Diagnostic of neurological disorder affecting central nervous system function
* Moderate to severe substance use disorders (>=4/11 as defined in DSM-5) and excluding smoking disorders
* Volunteers under court protection or guardianship
* Unable to give the volunteer informed information, or the volunteer refuses to sign the consent form
* Physiological condition deemed clinically incompatible with the study by the investigator o For subjects undergoing MRI: presence of a contraindication for MRI examination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Predictive value of ELK1 and GPR56 mRNA levels separately and in combination for the development of psychiatric symptoms following PTE at 6-month follow-up. | 6 months

SECONDARY OUTCOMES:
Predictive value of the resilience prognosis of a transcriptomic and epigenetic signature (non-coding RNAs and DNA methylation) including GPR56 and ELK1 non-exclusively for the appearance of psychiatric symptoms following a PTE | 12 months
Predictive value of structural MRI for the development of psychiatric symptoms following PTE | 12 months
  The AUC value determined by structural MRI prediction ROC curve analysis (morphometric analysis) for the onset of psychiatric symptoms during 6 and then 12 month follow-up period after PTE
Predictive value of measure of cognitive functioning for the development of psychiatric symptoms following PTE | 12 months
  The AUC value determined by ROC curve analysis of the MINI and WHODAS measure of cognitive functioning for the development of psychiatric symptoms at 6 and 12 month follow-up period after PTE.
Predictive value of transcriptomic and epigenetic signature for the development of psychiatric symptoms following PTE | 12 months
  The AUC value determined by ROC curve analysis of a transcriptomic and epigenetic signature predictive of the onset of psychiatric symptoms during 6 and then 12 month follow-up period after PTE
Predictive value of ELISA measurement of GPR56 and ELK1 in serum for the development of psychiatric symptoms following PTE | 12 months
  The AUC value determined by ROC curve analysis of the ELISA measurement of GPR56 and ELK1 in serum for the development of psychiatric symptoms during 6 and then 12 month follow-up period after PTE
Title: Predictive value of heart rate variability measuremen for the development of psychiatric symptoms following PTE | 12 months
  The AUC value determined by ROC curve analysis of the heart rate variability measurement for the onset of psychiatric symptoms during a 6- and then 12-month follow-up period after EFA.

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique Hopitaux De Marseille
Locations (4):
- France (4):
  - Hopital de la Conception, Marseille
  - Hopital Sainte Marguerite, Marseille
  - CHU Montpellier, Montpellier
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No